CLINICAL TRIAL: NCT05151419
Title: Comparative Study Between Endobronchial Forceps-Biopsy and Cryo-Biopsy in the Diagnosis of Bronchogenic Carcinoma
Brief Title: Forceps Biopsy Versus Cryo-biopsy in the Diagnosis of Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nashwa Ahmed Mohammad amin (Other)
Responsible Party: Sponsor-Investigator, Nashwa Ahmed Mohammad amin, Nashwa Ahmed Mohammad amin, Benha University
Organization: Benha University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21/7/2020
Record Dates: First submitted 2021-11-14; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Lung Cancer
Keywords: bronchoscope, cryo-biopsy
MeSH Terms: conditions — Lung Neoplasms | interventions — Bronchoscopes

STUDY DESIGN:
Intervention Model Description: A total number of 30 participants were enrolled in our study. These individuals had a diagnostic bronchoscopy because they had a suspicion of lung cancer and needed tissue samples to confirm the diagnosis. All of the procedures were carried out with 2% lidocaine instillation and midazolam IV sedation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bronchoscope ,forceps,cryo-biopsy (Other): biopies were taken from the lung mass using forceps and cryo-biopsy to evalute diagnostic yield of cryo-biosy versus forceps in the diagnosis of lung cancer
  Interventions: Procedure: bronchoscpe

INTERVENTIONS:
Procedure: bronchoscpe — bronchoscopic biopsy from lung mass using cryobiopsy and forceps
  Other Names: bronchoscope

SUMMARY:
This study was comprised of 30 patients who were scheduled for a diagnostic bronchoscopy due to a suspicion of lung cancer in order to obtain tissue samples for a final diagnosis , four biopsies were taken by each of cryobiopsy and forceps biopsy , to evaluate and compare the diagnostic yield of endobronchial cryobiopsy and forceps biopsy in the diagnosis of lung cancer .

DETAILED DESCRIPTION:
Diagnostic bronchoscopic interventions are used to evaluate and tissue sample from endobronchial lesions utilising variety of devices that can be delivered through the operative channel of a fibrio-optic bronchoscope.

All of the procedures were carried out with 2% lidocaine instillation and midazolam IV sedation All patients signed a written informed consent form for bronchoscopy and tissue sampling with forceps and a cryoprobe.between August 2020 and June 2021. All interventions were performed in the bronchoscopy unit of the Chest Medicine Department at Benha university Data were collected, revised, coded and entered to the Statistical Package for Social Science (IBM SPSS) version 23. The quantitative data with parametric distribution were presented as mean, standard deviations and ranges.

ELIGIBILITY:
Inclusion Criteria:

* severe uncorrected hypoxemia despite supplemental oxygen treatment
* unstable angina
* uncontrolled arrhythmias,
* severe hypercarbia,
* unstable cervical spine.
* Coagulopathy that cannot be reversed
* Chronic obstructive pulmonary disease (COPD) exacerbation
* Severe Illness
* old age
* malnutrition
* Patient who refused to have a bronchoscopy performed

Exclusion Criteria:

Patients' histories, including age, sex, and smoking status, were documented for all participants in the trial Clinical examination and medical history Complete blood count, serum creatinine, liver enzymes, INR, bleeding time, and clotting time are all routine laboratory tests Plain chest X-ray and chest computed tomography were used in the radiological workup* Arterial blood gas on room air. bronchoscopy and biopsy taking with forceps and cryobiopsy

-

Ages: 47 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2021-06-05 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
Comparative study between Endobronchial Forceps-Biopsy and Cryo-Biopsy in the Diagnosis of bronchogenic carcinoma | comprative , week 40
  The comparison between groups regarding qualitative data was done by using Chi-square test and/or Fisher exact test when the expected count in any cell found less than 5.at week 40

CONTACTS AND LOCATIONS:
Overall Officials: nashwa ah amin, MD, Principal Investigator — nashwa ahmed amin
Locations (1):
- Benha University Hospital- Chest Department, Cairo, Egypt